CLINICAL TRIAL: NCT00927667
Title: A Diagnostic Interventional, Controlled, Cross-sectional Evaluation of Joint Status Using Magnetic Resonance Imaging in Subjects With Severe Hemophilia A Treated With Primary Prophylaxis, Secondary Prophylaxis, or On-demand Therapy
Brief Title: Joint Status in Subjects With Severe Hemophilia A in Relation to Different Treatment Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare AG
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12948; 2009-010147-14 (EudraCT Number)
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Joint Status; Bleeds; Magnetic Resonce Imaging
MeSH Terms: conditions — Hemophilia A; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental)
  Interventions: Procedure: No Drug
- Arm 2 (Experimental)
  Interventions: Procedure: No Drug
- Arm 3 (Experimental)
  Interventions: Procedure: No Drug
- Arm 4 (Experimental)
  Interventions: Procedure: No Drug
- Arm 5 (Experimental)
  Interventions: Procedure: No Drug

INTERVENTIONS:
Procedure: No Drug — Patients have received primary FVIII prophylaxis (started < 2 years of age)
  Arms: Arm 1
Procedure: No Drug — Patients have received secondary FVIII prophylaxis (started 2 - < 6 years of age)
  Arms: Arm 2
Procedure: No Drug — Patients have received secondary FVIII prophylaxis (started 6 - < 12 years of age)
  Arms: Arm 3
Procedure: No Drug — Patients have received secondary VIII prophylaxis(started 12 - 18 years of age)
  Arms: Arm 4
Procedure: No Drug — Patients have received on-demand therapy
  Arms: Arm 5

SUMMARY:
The joint status (knees, ankles) of patients suffering from severe Hemophilia A (too little blood clotting factor VIII in blood) is evaluated in a single magnetic resonance imaging session. No study medication is given.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 12 - 35 years
* Severe hemophilia A ( < 1 % FVIII:C)
* No history of Factor VIII inhibitory antibody
* For prophylaxis groups, having received at least two prophylactic infusions per week for 45 weeks per year for the prevention of bleeding without relevant interruption and continuing until the present.
* Complete documentation of joints bleeds and their locations prior to start of prophylaxis,
* Bleeding history and/or treatments received during the last 5 years documented in the subjects medical records.
* For the on-demand subjects > 12 bleeds/year in the last 5 years.
* Written informed consent by subject and parent/legal representative, if < 18 years

Exclusion Criteria:

* Individuals with other coagulopathies (e.g., von Willebrand disease)
* HIV seropositive subjects
* Individuals for whom the most clinically severe joint is not one of the 4 index joints (ankle, knee)
* HCV seropositive individuals who underwent interferon therapy during the last 12 months
* Individuals for whom high-magnetic exposure is contraindicated (see section 7.1)
* Synovectomy performed within the six months prior to investigation enrollment or orthopedic surgery planned to be performed within the investigation period
* Joint replacement
* For the on-demand treatment group, any period greater than 8 consecutive months having received >/= 50 IU per kg per week Factor VIII for the prevention of bleeding

Ages: 12 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum ankle MRI score | no timeframe (single visit, "snapshot" of the actual joint status)

SECONDARY OUTCOMES:
Total MRI score of the maximum index joint | no timeframe (single visit, "snapshot" of the actual joint status)
Number of bleeds in each index joint over previous 5 years | no timeframe (medical history status)
Number of total joint bleeds and their locations over previous 5 years | no timeframe (medical history status)
Physical joint score (Gilbert Score) | no timeframe (single visit, "snapshot" of the actual joint status)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- Germany (4):
  - Heidelberg, Baden-Wurttemberg
  - Bonn, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Magdeburg, Saxony-Anhalt
- Athens, Greece
- Italy (4):
  - Milan
  - Padua
  - Parma
  - Roma
- Spain (2):
  - A Coruña, A Coruña
  - Valencia, Valencia
- Sweden (2):
  - Malmo
  - Stockholm
- United Kingdom (2):
  - Canterbury, Kent
  - London